CLINICAL TRIAL: NCT05505799
Title: Community Medical Center, Continuous Quality Improvement Project, Rapid Sequence Intubation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Community Medical Center, Toms River, NJ (Other)
Responsible Party: Principal Investigator, Greg Neyman, Sub-Investigator, Clinical Professor, Community Medical Center, Toms River, NJ
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 22-020
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-02

CONDITIONS: Intubation, Intratracheal; Rapid Sequence Induction and Intubation; Checklist
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Before and After study of a Checklist Intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preintervention (Active Comparator): Normal clinician intubation process
  Interventions: Other: Standard Care
- Postintervention (Experimental): Clinician intubation process after implementation and clinician education with a procedural checklist
  Interventions: Other: Intubation Checklist

INTERVENTIONS:
Other: Intubation Checklist — A preprocedure checklist will be made available to clinicians, and they will be educated on proper use of the checklist
  Arms: Postintervention
Other: Standard Care — Clinicians will intubate as per their usual practice
  Arms: Preintervention

SUMMARY:
To assess the ongoing continuous quality improvement of rapid sequence intubation in our emergency department. Ongoing assessment will address standardization of the process and protocol driven measures that will improve the overall quality of the intervention.

DETAILED DESCRIPTION:
Continuous evaluation and improvement of airway performance in the Emergency Department (ED) is essential for achieving positive clinical outcomes and reducing the incidence of related adverse events. First-pass success (FPS) in Rapid Sequence Intubation (RSI) is the most commonly utilized metric for evaluation and allows for comparison across clinical environments. According to a variety of studies published over the last decade, including a large, multi-center systematic review and meta-analysis, the mean FPS rate (84%) has been used as an institutional benchmark for ED airway proficiency.

Unfortunately, many complications can arise during RSI, the incidence of which has remained high. These complications commonly lead to poor or life-threatening outcomes and include desaturation, hypotension, dysrhythmia, cardiac arrest, pneumothorax, dental trauma, and esophageal intubation. According to the 4th National Audit Project of the Royal College of Anesthetists, it was determined that 30% of patients in the ED and 60% of patients in the ICU experiencing an airway related incident, suffered brain damage or death. The number of failed intubation attempts (3+) has been directly correlated with the an increased development of complications. Thus, establishing effective methods of decreasing the occurrence of failed attempts will result in an immediate reduction of unintended issues.

To maximize FPS and increase the safety of the procedure, it is essential to develop a tool to maximize efficacy. The introduction of checklists as a process improvement tool has been identified as a successful strategy for improving the effectiveness and quality of procedures throughout healthcare. Integration of a checklist in the RSI procedure will help to increase FPS rates and act as a method to aid in continuous evaluation and improvement of overall airway performance.

Although many airway performance improvement studies exist, our institution is unique in that we are a new Emergency Medicine (EM) Residency program that will be comprised of only post-graduate year 1 (PGY1) and post-graduate year 2 (PGY2) EM residents at the commencement of data collection. Furthermore, our clinical skills training process involves an integrative approach, pioneered by our interdisciplinary team of educators. Continuous evaluation of FPS and the incidence of RSI-related complications will allow for assessment of not only our quality improvement initiative, but of our educational methodology as well. Overall, implementation of quality and performance improvement strategies can mitigate the occurrence of adverse events and lead to improved health outcomes for our patients. This is of paramount importance to us as providers and to our community as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Any patient undergoing endotracheal intubation in the Emergency department

Exclusion Criteria:

* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
First Pass Success Rate | At time of intubation
  Proportion of intubations where the trachea is successfully intubated on the first attempt

SECONDARY OUTCOMES:
Aspiration rate | At time of intubation
  Proportion of intubations where patients suffer aspiration
Cardiac arrest | At time of intubation
  Proportion of intubations where patients suffer cardiac arrest
Cuff Leak | At time of intubation
  Proportion of intubations where the endotracheal tube experiences a cuff leak
Dental trauma | At time of intubation
  Proportion of intubations where patients suffer dental trauma
Dysrhythmia | At time of intubation
  Proportion of intubations where patients suffer dysrhythmia
Esophageal intubation | At time of intubation
  Proportion of intubations where patients encounter esophageal intubation
Unplanned extubation | At time of intubation
  Proportion of intubations where patients encounter an unplanned extubation
Post procedural hypotension | At time of intubation
  Proportion of intubations where patients suffer hypotension in the immediate postprocedure period
Hypoxemia | At time of intubation
  Proportion of intubations where patients suffer hypoxemia
Laryngospasm | At time of intubation
  Proportion of intubations where patients suffer laryngospasm
Mainstem intubation | At time of intubation
  Proportion of intubations where patients encounter a mainstem intubation

CONTACTS AND LOCATIONS:
Overall Officials: Josesph Roarty, MD, Principal Investigator — Robert Wood Johnson Barnabas Health Community Medical Center
Locations (1):
- Community Medical Center, Toms River, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakles JC, Augustinovich CC, Patanwala AE, Pacheco GS, Mosier JM. Improvement in the Safety of Rapid Sequence Intubation in the Emergency Department with the Use of an Airway Continuous Quality Improvement Program. West J Emerg Med. 2019 Jul;20(4):610-618. doi: 10.5811/westjem.2019.4.42343. Epub 2019 Jun 3. PMID 31316700
- [Background] Turner JS, Bucca AW, Propst SL, Ellender TJ, Sarmiento EJ, Menard LM, Hunter BR. Association of Checklist Use in Endotracheal Intubation With Clinically Important Outcomes: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Jul 1;3(7):e209278. doi: 10.1001/jamanetworkopen.2020.9278. PMID 32614424
- [Background] Park L, Zeng I, Brainard A. Systematic review and meta-analysis of first-pass success rates in emergency department intubation: Creating a benchmark for emergency airway care. Emerg Med Australas. 2017 Feb;29(1):40-47. doi: 10.1111/1742-6723.12704. Epub 2016 Oct 27. PMID 27785883
- [Background] Sakles JC, Chiu S, Mosier J, Walker C, Stolz U. The importance of first pass success when performing orotracheal intubation in the emergency department. Acad Emerg Med. 2013 Jan;20(1):71-8. doi: 10.1111/acem.12055. PMID 23574475
- [Background] Bernhard M, Becker TK, Gries A, Knapp J, Wenzel V. The First Shot Is Often the Best Shot: First-Pass Intubation Success in Emergency Airway Management. Anesth Analg. 2015 Nov;121(5):1389-93. doi: 10.1213/ANE.0000000000000891. No abstract available. PMID 26484464
- [Background] Sakles JC, Mosier JM, Patanwala AE, Arcaris B, Dicken JM. First Pass Success Without Hypoxemia Is Increased With the Use of Apneic Oxygenation During Rapid Sequence Intubation in the Emergency Department. Acad Emerg Med. 2016 Jun;23(6):703-10. doi: 10.1111/acem.12931. Epub 2016 May 13. PMID 26836712
- [Background] Gopinath B, Sachdeva S, Kumar A, Kumar G. Advancing emergency airway management by reducing intubation time at a high-volume academic emergency department. BMJ Open Qual. 2021 Jul;10(Suppl 1):e001448. doi: 10.1136/bmjoq-2021-001448. PMID 34344738
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948